CLINICAL TRIAL: NCT06523257
Title: Prevalence of Chronic Obstructive Pulmonary Disease in the Portuguese Population- EpiCOPDpt Study
Brief Title: Prevalence of Chronic Obstructive Pulmonary Disease in the Portuguese Population
Acronym: EpiCOPDpt
Status: Not yet recruiting | Type: Observational
Sponsor: Sociedade Portuguesa de Pneumologia (Other)
Responsible Party: Sponsor
Other Study IDs: 2023_EO_EPICOPDPT
Record Dates: First submitted 2024-07-16; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Spirometry

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Spirometry — Spirometry is a simple test used to diagnose and monitor lung diseases by measuring how much air a person can breathe out in one forced breath.
  After the baseline spirometry, and only if there is clear evidence of an airflow limitation/obstruction, i.e., if the FEV1/FVC (forced expiratory volume in the first second/forced vital capacity) ratio is less than 70% or less than the 5th percentile of the distribution of values measured in the reference population, a bronchodilator test will be performed using standardised post-bronchodilator spirometry (200 µg salbutamol), in order to identify persistent airflow limitation/obstruction.

SUMMARY:
The EpiCOPDpt Study (Prevalence of Chronic Obstructive Pulmonary Disease in the Portuguese Population) primary objective is to estimate the prevalence of Chronic Obstructive Pulmonary Disease (COPD) in the Portuguese population aged 20 and over. It is a cross-sectional study of a representative sample of the Portuguese population aged 20 and over, using standardised post-bronchodilator spirometry. Questionnaires will be applied to collect sociodemographic, economic, clinical, and therapeutic data.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 20 years and over, with permanent or temporary residence for at least one year in the national territory;
* Written informed consent for study participation.

Exclusion Criteria:

* Any condition that makes it impossible to perform spirometry, in accordance with standards of the joint American Thoracic Society/European Respiratory Society, and as described in the "Contraindications for spirometry testing" section of the Study Procedures Manual;
* Any condition that makes it impossible to perform the bronchodilation, as described in the "Contraindications for bronchodilation" section of the Study Procedures Manual;
* Severe cognitive disability that may interfere with the person's capability to participate in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Portuguese population aged 20 years and over.
Sampling Method: Probability Sample
Enrollment: 8589 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Individuals aged 20 years and over in the Portuguese population diagnosed with COPD(Chronic Obstructive Pulmonary Disease). | Through study completion, an average of 10 months
  Number and proportion of individuals aged 20 years and over in the Portuguese population diagnosed with COPD.

SECONDARY OUTCOMES:
Individuals aged 20 years and over in the Portuguese population diagnosed with COPD (Chronic Obstructive Pulmonary Disease), by age group | Through study completion, an average of 10 months
  Number and proportion of individuals aged 20 years and over in the Portuguese population diagnosed with COPD among males and females, within specific age groups (≥20, 20-29, 30-39, 40-49, 50-59, 60-69, and ≥70).
Individuals aged >20 years in the Portuguese population diagnosed with COPD (Chronic Obstructive Pulmonary Disease) by sex | Through study completion, an average of 10 months
  Number and proportion of individuals aged 20 years and over in the Portuguese population diagnosed with COPD by sex: males and females.
Individuals diagnosed with COPD (Chronic Obstructive Pulmonary Disease) in each NUTS region | Through study completion, an average of 10 months
  Number and proportion of individuals diagnosed with COPD in each NUTS region (Norte, Centro, Lisboa e Vale do Tejo, Alentejo, Algarve, Açores, and Madeira).
Sociodemographic profile of respiratory patients | Through study completion, an average of 10 months
  A set of characteristics will be used to determine the sociodemographic profile: Sociodemographic characteristics:
  * Age
  * Sex
  * Race
  * Ethnicity
  * Marital status
  * Education level
  * Socioeconomic status (income and living conditions) Number and proportion in case of categorical data and means, std dev and percentiles in case of continuous variables.
Clinical profile of respiratory patients | Through study completion, an average of 10 months
  A set of characteristics will be used to determine the clinical profile:
  * Respiratory symptoms (such as cough, shortness of breath, and wheezing)
  * Comorbidities (Yes, which?/No)
  * Lung function tests (Spirometry will be carried out in accordance with the standard protocol of the joint ATS/ERS. The US Third National Health and Nutrition Examination Survey (NHANES III) values will be used as reference. Peripheral blood oxygen saturation (SpO2) will be assessed using a pulse oximeter)
  * Anthropometric data: Weight in kilograms and height in meters. Weight and height will be combined to report BMI in kg/m^2.
  Number and proportion in case of categorical data and means, std dev and percentiles in case of continuous variables.
Risk profile of participants | Through study completion, an average of 10 months
  Characterisation of risk factors, such as smoking history, occupational exposures, air pollution exposure, genetic predisposition, and history of respiratory infections. Number and proportion in case of categorical data and mean, median, standard deviation, and percentiles in case of continuous variables.

IPD SHARING:
Plan to Share IPD: Undecided